CLINICAL TRIAL: NCT02909075
Title: An Initial Study of FDG-PET/CT and MRI to Assess Thymic Function
Brief Title: A Study to Assess Thymic Function Using PET/CT and MRI
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1244
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: CD34 Selected Peripheral Blood Stem Cell Graft
Keywords: PET/CT; MRI; Assess Thymic Function; 16-1244
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- PET/CT scans and MRI: Eligible patients will be enrolled onto the study, and will undergo 3 limited field of view (FOV) FDG-PET/CT scans and MRI of the chest: at baseline (within 4 weeks prior to transplantation), and approximately 3 months (+/-2 weeks) and 6 months (+/-2 weeks) after transplant. PET/CT and MR imaging can be completed on the same day. We will also offer the exams on other days if this is easier for the patient. The PET/CT and MR should be performed within 2 weeks of each other.
  Interventions: Device: PET/CT scans; Device: MRI

INTERVENTIONS:
Device: PET/CT scans
Device: MRI

SUMMARY:
The purpose of this study is to see if a positron emission tomography/computed tomography (PET/CT) scan and a magnetic resonance imaging (MRI) of the chest can assess changes in the thymus size and function. The researchers would like to monitor the thymus with a PET/CT scan and a MRI before and after the participants transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age is ≥18 or ≤65 years old.
* Patients must have a plan to receive a CD34-selected peripheral blood stem cell graft.

Exclusion Criteria:

* Patient is not able to undergo MR imaging due to any contraindication to MRI based on departmental MR questionnaire (e.g. past gadolinium allergies, failure of metallic screening, claustrophobia, inability to lay flat for duration of the study, inability to hold breath, etc.)
* Pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSK BMT clinic
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-08; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
change in thymic size | 1 year
  A clinically meaningful change is defined as increase in thymic size (> 0.2cm increase in uni-dimensional diameter), functional volume (>10%) or uptake (≥25%). We will report proportion of patients with each component of clinically meaningful change, as well as the proportion with at least one component, along 95% exact confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schoder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/